## INFORMED CONSENT FORM

(For Control Group)

This study is carried out as a master's thesis under the supervision of Assistant professor Semra ÇEVİK by Serap KARADUMAN from Gaziantep University Faculty of Health Sciences. The study was planned to determine the effect of massage applied during labor on the woman's fear, anxiety and perception of labor pain. No other treatment or treatment will be done to you during the research. Only at different times by the researcher you will be asked some survey questions and your answers will be recorded. The data will be used for scientific purposes and the individual data will be kept confidential.

Thank you.

Serap KARADUMAN

Gaziantep University Faculty of Health Sciences

Date Signature

## INFORMED CONSENT FORM

(For Experimental Group)

This study is carried out as a master's thesis under the supervision of Assistant professor Semra ÇEVİK by Serap KARADUMAN from Gaziantep University Faculty of Health Sciences. The study was planned to determine the effect of massage applied during labor on the woman's fear, anxiety and perception of labor pain. Massage will be applied to your sacral region. The application of the massage will be applied during the birth pains and will be continued for 30 minutes in each application. No discomfort will be felt during all these applications. At different times the researcher will ask you some questionnaire questions and your answers will be recorded. You have the right to learn all the information you need and ask questions. The application of massage to the sacral region has no detrimental effect on health.



The data will be used for scientific purposes and the individual data will be kept confidential. Thank you.

## Serap KARADUMAN

Gaziantep University Faculty of Health Sciences

| I, | |
|---|---|
| above. I v | was informed orally about the research. I agree to participate in the research at any |
| stage of t | he research without affecting the service provided to me. |

Date Signature